CLINICAL TRIAL: NCT04239040
Title: A Phase 1 Study of Combination Nivolumab and Ipilimumab With Irradiated GM-CSF Secreting Autologous Neuroblastoma Cell Vaccine (GVAX) for Relapsed or Refractory Neuroblastoma
Brief Title: GVAX Plus Checkpoint Blockade in Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Manufacturing issues
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Natalie Collins, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-680
Record Dates: First submitted 2020-01-21; First posted 2020-01-23 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Neuroblastoma; Pediatric Solid Tumor
Keywords: Neuroblastoma; Pediatric Solid Tumor; Immunotherapy; GVAX Vaccine; Nivolumab; Ipilimumab
MeSH Terms: conditions — Neuroblastoma | interventions — Tissue Banks; GVAX vaccine; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relapsed or Refractory High Risk Neuroblastoma (Experimental): Tissue Collection of Cancerous cells during primary or clinically indicated surgical resection.
  Manufacture and cryopreservation of vaccine. Treatment with vaccine, nivolumab and ipilimumab.
  * Vaccine injected weekly over initial 21 day cycle, biweekly for cycles 2-4 of 21 day cycle duration and cycles 5 and subsequent of 28 day cycle duration until vaccine supply is exhausted.
  * Intravenous infusion of nivolumab every 3 weeks, for cycles 1-4. Cycles 1-4 are 21 days
  * Intravenous infusion of ipilimumab every 3 weeks, for cycles 1-4. Cycles 1-4 are 21 days
  * Intravenous infusion of nivolumab biweekly for cycle 5 and subsequent of 28 day cycle duration. Subsequent 28 day cycles will last up to 2 years.
  Interventions: Procedure: Tissue collection; Biological: GVAX vaccine; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Procedure: Tissue collection — Collection of cancerous tissue to create GVAX vaccine or irradiated GMCSF-secreting autologous neuroblastoma cell vaccine at time of clinically indicated surgical procedure
Biological: GVAX vaccine — Vaccine injected weekly over initial 21 day cycle, biweekly for cycles 2-4 of 21 day cycle duration and cycles 5 and subsequent of 28 day cycle duration until vaccine supply is exhausted.
  Other Names: GMCSF-secreting autologous neuroblastoma cell vaccine
Drug: Nivolumab — Intravenous infusion of nivolumab every 3 weeks, for cycles 1-4. Cycles 1-4 are 21 days
  Intravenous infusion of nivolumab biweekly for cycle 5 and subsequent of 28 day cycle duration. Subsequent 28 day cycles will last up to 2 years.
  Other Names: Opdivo
Drug: Ipilimumab — Intravenous infusion of ipilimumab every 3 weeks, for cycles 1-4. Cycles 1-4 are 21 days
  Other Names: Yervoy

SUMMARY:
This research clinical trial is studying the creation and administration of GVAX, an irradiated GM-CSF secreting, autologous neuroblastoma cell vaccine (GVAX) in combination with nivolumab and ipilimumab as a possible treatment for neuroblastoma.

The names of the study drugs involved in this study are:

* GVAX Vaccine, an immunotherapy developed from surgically removed tumor tissue
* Nivolumab
* Ipilimumab

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved the GVAX vaccine as a treatment for any disease.

The U.S. Food and Drug Administration (FDA) has not approved nivolumab or ipilimumab for your specific disease but it has been approved for other uses.

The research study procedures include: screening for eligibility and study treatment including evaluations and follow up visits.

This phase 1 study will be conducted in 2 parts

* In the first part, participants will, as part of standard of care procedure to remove cancerous tissue, undergo neuroblastoma cell collection from a portion of resected tumor.
* Those cells will then be used to create the vaccine which will be stored for potential use during the second part of this research study.
* In the second part, participants who did not respond to standard therapy will receive the GVAX vaccine along with nivolumab and ipilimumab.

The study treatment will continue for up to 24 months and participants will be followed for 2 years after last study treatment (if received at least one vaccination).

ELIGIBILITY:
Inclusion Criteria:

* Eligibility Criteria for neuroblastoma cell collection and vaccine manufacture

  * Patients with histologically confirmed neuroblastoma, who meet the Children's Oncology Group (COG) high-risk group assignment criteria
  * Lansky/Karnofsky performance status ≥50% (see Appendix A)
  * Participants must have clinical indication for surgical resection of their neuroblastoma and undergo resection at Boston Children's Hospital
  * Ability to understand and/or the willingness of their parent or legally authorized representative to sign a written informed consent document.
* Eligibility Criteria to commence to receive study treatment with irradiated GM-CSF secreting autologous tumor vaccine, nivolumab, and ipilimumab

  * Histologically confirmed high-risk neuroblastoma based on COG assignment criteria
  * Residual disease at the end of standard therapy or relapsed neuroblastoma in any disease state (including CR) by clinical criteria (histologic confirmation of relapse or residual disease is not required).
  * Age > 1 year of age
  * Lansky/Karnofsky performance status ≥50% (see Appendix A)
  * Prior Therapy - Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimal duration from prior anti-cancer directed therapy prior to enrollment

    * Myelosuppressive Chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy
    * Small molecule biologic therapy: At least 7 days following the last dose of a biologic agent.
    * Monoclonal antibodies ≥ 7 days or 3 half-lives whichever is longer but no longer than 30 days (with recovery of any associated toxicities)
    * External beam irradiation: ≥ 14 days after small port XRT, ≥ 12 weeks after large port radiation (≥ 50% of the marrow space) including total body irradiation, craniospinal radiation, whole abdomen and whole lung radiation
    * 131I- MIBG therapy ≥ 6 weeks
    * Autologous stem cell infusion following myeloablative therapy ≥ 6 weeks
    * Any other investigational agents ≥ 14 days
* Organ function requirements

  * Adequate bone marrow function defined as:

    * ANC >/= 500/µL
    * Hgb >8 (may not be transfused)
    * Platelet count ≥30,000 (may not be transfused)
  * Hepatic Function:

    * Total bilirubin ≤ 1.5 x upper limit of normal for age
    * ALT (SGPT) ≤ 3 x upper limit of normal (135 U/L) For the purpose of this study, the ULN for ALT is 45 U/L
  * Renal Function, a serum creatinine based on age/sex as follows:

    * Maximum Serum Creatinine (mg/dL)

      * Age 1 to <2 years Male: 0.6 Female: 0.6
      * Age 2 to < 6 years Male:0.8 Female 0.8
      * Age 6 to < 10 years Male:1 Female: 1
      * Age 10 to < 13 years Male: 1.2 Female: 1.2
      * Age 13 to < 16 years Male: 1.5 Female: 1.4
      * Age ≥ 16 years Male: 1.7 Female: 1.4
    * OR Creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels greater than the above age/sex maximum allowed values
  * Adequate Pulmonary Function Defined as:

    * No evidence of dyspnea at rest
    * No exercise intolerance due to pulmonary insufficiency
    * Pulse oximetry > 92% while breathing room air
  * Adequate pancreatic function defined as

    * Serum lipase </= ULN at baseline.
  * No ≥ Grade 2 non-hematologic toxicity
  * Absolute eosinophil count ≤ 5000/ul
  * Negative B-HCG pregnancy test in females of childbearing potential. Must be drawn or repeated within 24 hours prior to initial administration of study drugs
  * Women of childbearing potential (WOCBP) receiving nivolumab will be agree to adhere to contraception for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are sexually active with WOCBP will agree to adhere to contraception for a period of 7 months after the last dose of nivolumab.

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* No systemic corticosteroid therapy, other than replacement therapy for adrenal insufficiency or transfusion premedication. Participants who are receiving or have received lympholytic steroid (>=40mg/m2 prednisone equivalent) therapy within 4 weeks of first anticipated vaccine administration are excluded, because high-dose steroid therapy is expected to significantly limit the ability of the immune system to respond to GVAX vaccination.
* Participants with known parenchymal brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GM-CSF or DMSO.
* Participants with any form of primary immunodeficiency.
* Females who are pregnant are excluded from this study because GVAX is an investigational biologic with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with GVAX, breastfeeding should be discontinued if the mother is treated with GVAX
* Uncontrolled intercurrent illness or serious uncontrolled medical disorder including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia and/or pronounced disturbances of the electrical conduction system of the heart or psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV-positive participants on combination antiretroviral therapy are ineligible because of the effect of GVAX vaccination on the disease course is unknown and because the underlying disease is expected to limit the ability of the immune system to respond to GVAX vaccination.
* Clinically relevant known active infection including active hepatitis B or C or any other concurrent disease which in the judgment of the Investigator would make the subject inappropriate for enrollment on this study
* History of a malignancy other than neuroblastoma with exception of the following circumstances:

  * Patients with a history of malignancy who have been adequately treated and have been disease-free for at least 2 years are not excluded.
  * Patients with adequately treated active non-invasive cancers (such as non-melanomatous skin cancer or in-situ bladder, cervical and breast cancers) are not excluded.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti PD L2 or anti-CTLA4 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. OX 40, CD137).
* Has active autoimmune disease that has required systemic treatment in the past 12 months, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy are exceptions. Intermittent use of bronchodilators or local steroid injections are not excluded. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Autoimmune diagnoses not listed must be approved by the protocol chair.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
The number of participants with grade 4 toxicities | Up to 2 years
  To assess safety, the number of grade 4 toxicities associated with vaccine and nivolumab/ipilimumab using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5
Number of Participants to receive 6 vaccinations | Up to 2 years
  Feasibility will be assessed by the ability to make vaccine from available biopsy material in quantities sufficient for six vaccinations, for a given patient. A success rate (number of patients for whom quantity sufficient for six vaccinations exist / total number of eligible patients) under 65% may imply that the method needs further development or that the amount of tissue available in this population limits the feasibility of this strategy. Total number of vaccine doses administered per patient will also be counted

SECONDARY OUTCOMES:
Progression-free survival (PFS) | time from receipt of first GVAX vaccine dose to the earlier of progression, relapse or death due to disease up to 48 months
  Kaplan-Meier plots, 1-year PFS estimate will be calculated, along with the standard errors
Overall best response | Start of the treatment until disease progression/recurrence up to 48 months
  Each patient will be categorized as a responder (≥PR) or a non-responder (<PR) by INRC criteria
Overall Survival | Time from receipt of the first GVAX vaccine dose to death due to any cause up to 48 months
  Kaplan-Meier plots, 1-year OS estimates will be calculated, along with the standard errors

CONTACTS AND LOCATIONS:
Overall Officials: Natalie B Collins, MD, PHD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institite, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu